CLINICAL TRIAL: NCT05407870
Title: A Comparative Study of the Efficacy and Safety of Etomidate Compared to Propofol in Gastric Endoscopic Submucosal Dissection: a Prospective, Single-center, Randomized, Double-blind, Non-inferiority Study
Brief Title: Efficacy and Safety of Etomidate Sedation in Gastric Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Keum, Bo Ra, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020AN0375
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Sedation Complication; Endoscopic Submucosal Dissection; Esophagogastroduodenoscopy
Keywords: Etomidate; Propofol
MeSH Terms: interventions — Etomidate; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator): induction - 0.5mg/kg Propofol maintenance - 0.25mg/kg Propofol
  Interventions: Drug: Propofol Injection
- Etomidate (Experimental): induction - 0.25mg/kg Propofol + 0.05mg/kg Etomidate maintenance - 0.05mg/kg Etomidate
  Interventions: Drug: Etomidate Injection

INTERVENTIONS:
Drug: Etomidate Injection — Proofol and etomidate are drugs used for sedation and have the same white color.
  Gastric endoscopic submucosal dissection is performed using propofol in the control group and etomidate in the experimental group.
  Efficacy and safety of sedatives were confirmed using propofol and etomidate.
  Arms: Etomidate
Drug: Propofol Injection — Proofol and etomidate are drugs used for sedation and have the same white color.
  Gastric endoscopic submucosal dissection is performed using propofol in the control group and etomidate in the experimental group.
  Efficacy and safety of sedatives were confirmed using propofol and etomidate.
  Arms: Propofol

SUMMARY:
During endoscopy, the patient is sedated to relieve pain and improve the ease of the procedure. Sedation endoscopy using propofol is effective, but has the disadvantage that cardiopulmonary side effects are frequently observed. However, etomidate is known to have hemodynamic and respiratory stability.The purpose of this study was to compare the efficacy and safety of etomidate and propofol in sedated gastric endoscopic submucosal dissection.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80
* American Society of Anesthesiologists Physical Status Classification System (ASA) score of I, II, III
* Scheduled endoscopy

Exclusion Criteria:

* Pregnancy
* Previous study History of hypersensitivity to drugs or substances containing soy or egg ingredients
* Those who think that tracheal intubation will be difficult
* Obstructive sleep apnea
* History of side effects from previous sedatives
* People with severe liver disease, kidney disease, or heart disease
* Those who want a non-sleeping endoscope
* A person who refuses to provide consent
* SBP < 80mmHg or SpO2 < 90%
* Patients with adrenocortical dysfunction, chronic steroid users

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Respiratory adverse event | during gastric endoscopic submucosal dissection
  the number and proportion of cases of respiratory depression

SECONDARY OUTCOMES:
ESD clinical outcomes | From enrollment to the first clinic visit (within 60 days)
  tumor location, tumor pathology, ESD specimen size, En-bloc resection, submucosal invasion, margin positive
Adverse events and procedure interruptions | during gastric endoscopic submucosal dissection
  Overall adverse events Cardiopulmonary adverse events Procedure-related adverse events
  Overall procedure interruption procedure interruption due to cardiopulmonary adverse events procedure interruption due to procedure-related adverse events
Sedation-related profile | From initial administering the sedative drug to endoscopy room discharge (up to 2 hours); dose (ml)
  administered dose of sedatives (induction dose, maintenance dose, total dose), induction time, awake time, sedation time
Satisfaction assessment | From initial administering the sedative drug to endoscopy room discharge; satisfaction score (0-10, 10 is the highest score)
  patient satisfaction regarding sedation, doctor and nurse satisfaction regarding sedation during ESD
Hemodynamic changes | From date of randomization until the date of first documented progression (up to 2 hours)
  systolic blood pressure, diastolic blood pressure, mean arterial blood pressure, heart rate, oxygen saturation
Factors associated with adverse events | From date of randomization until the date of first documented progression (up to three days)
  factor analysis regarding overall adverse events factor analysis regarding overall cardiopulmonary adverse events factor analysis regarding overall procedure adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, Seoung-buk Gu, South Korea

IPD SHARING:
Plan to Share IPD: No